CLINICAL TRIAL: NCT01760252
Title: Neoadjuvant CAPOXIRI Chemotherapy in the Treatment of Resectable, Borderline Resectable and Locally Advanced Pancreatic Adenocarcinoma Protocol
Brief Title: Neoadjuvant CAPOXIRI Chemotherapy in the Treatment of Pancreatic Adenocarcinoma Protocol
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Medical Center (Other)
Collaborators: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CAPOXIRI
Record Dates: First submitted 2012-05-18; First posted 2013-01-04 (Estimated); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Metastatic Pancreatic Adenocarcinoma
Keywords: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Capecitabine; Oxaliplatin; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CAPOXIRI Chemotherapy Regimen (Experimental): Capecitabine, Oxaliplatin and Irinotecan (CAPOXIRI)
  The proposed chemotherapy regimen CAPOXIRI is:
  * Capecitabine 1000mg/m2 p.o. bid on days 1-7
  * Oxaliplatin 85mg/m2 intravenously (IV) on day 1
  * Irinotecan 150mg/m2 IV on day 1
  Interventions: Drug: Capecitabine, Oxaliplatin and Irinotecan (CAPOXIRI)

INTERVENTIONS:
Drug: Capecitabine, Oxaliplatin and Irinotecan (CAPOXIRI) — Neoadjuvant CAPOXIRI chemotherapy is an innovative strategy that builds on the advancement associated with FOLFIRINOX chemotherapy in patients with metastatic disease

SUMMARY:
The combination of capecitabine, oxaliplatin, and irinotecan (CAPOXIRI) may be better than other combinations used to treat earlier stage pancreatic cancer patients with resectable (able to be cut out), borderline resectable, and locally advanced pancreatic adenocarcinoma. For subjects who can not obtain Capecitabine can be treated with 5-Fluorouracil (5-FU) along with Oxaliplatin and Irinotecan. Though all of the drugs in this study have been approved by the FDA, their combination is investigational. The purpose of this study is to evaluate the effects of CAPOXIRI (good and bad) on you and your cancer.

DETAILED DESCRIPTION:
Introduction:

This is a phase II study evaluating the treatment adherence rate, efficacy and safety of neoadjuvant chemotherapy with capecitabine, oxaliplatin and irinotecan (CAPOXIRI) in patients with resectable (able to be cut out), borderline resectable and locally advanced pancreatic adenocarcinoma. Neoadjuvant CAPOXIRI chemotherapy is an innovative strategy that builds on the advancement associated with oxaliplatin, irinotecan, fluorouracil, and folinate (FOLFIRINOX regimen) chemotherapy in patients with metastatic disease. Building on the FOLFIRINOX regimen the use of CAPOXIRI is among the most clinically relevant projects for patients diagnosed with earlier stage pancreatic adenocarcinoma with the goal of improving patient outcomes and advancing our knowledge and understanding of this devastating disease.

The primary end point is the treatment adherence rate (TAR) which is the percentage of patients who complete 75% of the planned treatment (dose) for their diagnostic strata (resectable disease and borderline resectable/locally advanced disease).

Secondary end points are: Overall survival (OS), Disease-free survival (DFS; for those patients who are rendered disease-free by surgical resection), Progression Free Survival (PFS), Response Rate (RR), toxicity, and R0 resection rate (for patients stratified as having resectable disease and borderline resectable disease).

Background and Study Rationale:

It is estimated that 36,800 people will die of pancreatic cancer in the United States in 2010. Surgical resection offers the only chance of cure, but only 15-20% of cases are potentially resectable at present. Furthermore, prognosis is poor, even for those undergoing complete resection. Reported five-year survival rates following pancreatic-duodenectomy (surgery of the small intestine and pancreas) for node-negative disease is 25-30% and for node-positive disease is 10%.

The purpose of this study is to evaluate the effects of the combination of capecitabine, oxaliplatin, and irinotecan (CAPOXIRI) on the disease. This research is being done because we think that this combination, CAPOXIRI, may be better than other combinations used to treat your stage of pancreatic cancer.

A research study like this one has been done which shows that a similar combination of drugs including oxaliplatin, irinotecan and 5-fluorouracil (which is in the same class as capecitabine) can be effective in treating patients with pancreatic cancer who have more advanced disease than you. All of the drugs that are being used in this study have been approved by the FDA (Food and Drug Administration).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of pancreatic adenocarcinoma that is clinically staged as resectable, borderline resectable, or locally advanced as determined by CT criteria.
2. Age ≥ 18 years old.
3. An Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2 (Appendix B).
4. Patients must give written informed consent as per institutional and federal regulatory requirements.
5. An interval between initial diagnosis and consent of ≤ 42 days.
6. An interval between consent and initiating protocol-directed therapy of ≤ 14 days.
7. CT scan to stratify as resectable versus borderline resectable/locally advanced status within 28 days of initiating protocol-directed therapy.
8. A general level of health that would indicate a life expectancy of 5 years, excluding the patient's cancer diagnosis.
9. No prior chemotherapy, immunotherapy or radiotherapy for pancreatic adenocarcinoma.
10. Patients must have measurable or evaluable disease by Response Evaluation Criteria in Solid Tumors (RECIST) criteria (Appendix C).
11. Absolute granulocyte count of ≥ 1,500/mm3 and a platelet count of ≥ 100,000/mm3.
12. Patients must have adequate liver and renal function defined by a bilirubin of ≤ 2.0 mg/dL (with or without biliary stenting) and a creatinine of ≤ 1.5 mg/dL respectively.
13. Men and women who are fertile must use adequate contraception. Premenopausal women must have a negative pregnancy test documented prior to study entry.
14. There must be no extra-pancreatic spread of disease.
15. Patients must not have other serious illness or medical conditions including, but not limited to the following: New York Heart Association (NYHA) Class II or greater congestive heart failure or unstable angina pectoris, uncontrolled hypertension or arrhythmias, active bacterial infections, or unstable diabetes mellitus.
16. Patients must be disease-free of prior invasive malignancies for ≥ 5 years with the exception of curatively-treated basal cell or squamous cell carcinoma of the skin.

Exclusion Criteria:

1. Patients less than 18 years of age.
2. CT evidence of metastatic disease.
3. Pregnancy or considering pregnancy at the time of study entry.
4. Breast feeding at the time of study entry.
5. Prior therapy for pancreatic cancer including irradiation, chemotherapy, or immunotherapy.
6. Receiving concurrent chemotherapy, immunotherapy, or radiotherapy that is not part of this protocol while participating in this study.
7. Receiving concurrent treatment with any other investigational drug while on this protocol.
8. Prior malignancy within 5 years, excluding squamous or basal cell carcinoma of the skin that has been effectively treated, carcinoma in situ of the cervix, lobular carcinoma in situ of the breast, or ductal carcinoma in situ of the breast.
9. Non-malignant disease that would preclude protocol participation or follow-up.
10. Myocardial infarction within 6 months before enrollment, New York Heart Association (NYHA) Class II or greater heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, clinically significant pericardial disease, or electrocardiographic evidence of acute ischemic or active conduction system abnormalities.
11. Psychiatric disorders or conditions, that in the opinion of the investigator, would preclude the patient from providing truly informed consent.
12. Presence of progressive sensory neuropathy or progressive hearing loss or tinnitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-12; Primary Completion 2018-02-21 (Actual); Study Completion 2018-02-21 (Actual)

PRIMARY OUTCOMES:
The primary end point is the treatment adherence rate (TAR) which is the percentage of patients who complete 75% of the planned treatment (dose) for their diagnostic strata (resectable disease and borderline resectable/locally advanced disease) | 5 years
  Adherence of subjects with treatment

SECONDARY OUTCOMES:
Overall survival (OS), | 5 years
Progression Free Survival (PFS), | 5 years
Response Rate (RR), | 1 year
R0 resection rate for patients stratified as having resectable disease and borderline resectable disease. | 5 years
Disease-free survival (DFS; for those patients who are rendered disease-free by surgical resection), | 5 year

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kozuch, MD, Principal Investigator — Beth Israel Medical Center
Locations (3):
- United States (3):
  - Mount Sinai Beth Israel, New York, New York
  - St-Lukes Roosevelt Hospital Medical Center, New York, New York
  - Beth Israel Comprehensive Care Center, New York, New York